CLINICAL TRIAL: NCT01729832
Title: Intraoperative Stereotactic Image-guided Navigation of Perforators for DIEP Flap Breast Reconstruction.
Brief Title: Stereotactic Image-Guided Navigation During Breast Reconstruction in Patients With Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-10106; NCI-2012-00693 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (image-guided breast reconstruction) (Experimental): Patients undergo DIEP flap breast reconstruction using the StealthStation navigation system.
  Interventions: Procedure: breast reconstruction; Procedure: intraoperative imaging

INTERVENTIONS:
Procedure: breast reconstruction — Undergo DIEP flap breast reconstruction using the StealthStation navigation system
  Other Names: Mammaplasty
Procedure: intraoperative imaging — Undergo DIEP flap breast reconstruction using the StealthStation navigation system

SUMMARY:
Many hospitals, including the Ohio State University Medical Center, will take pictures of the blood vessels in a patient's abdomen before they decide to perform a breast reconstruction using the patient's own tissue. These pictures are called computed tomography (CT) angiograms and are like a map of each patient's anatomy. However, no study has been reported that determined how accurate these pictures are at showing the surgeon where all of the blood vessels were located. This study will try to determine if these pictures are missing any blood vessels that are found during surgery and if the pictures show the correct location of the vessels

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To analyze the accuracy of preoperative CT angiography in determining the location of perforator vessels. Through the use of an intraoperative navigation system, we will objectively locate perforators during surgery and compare the results to the preoperative imaging assessment of the flap's vascular anatomy.

II. To determine whether the preoperative CT angiogram allows the microsurgeon to correctly identify the perforators that are ultimately used as the pedicle for the flap.

OUTLINE:

Patients undergo deep inferior epigastric perforator (DIEP) flap breast reconstruction using the StealthStation navigation system.

After completion of study treatment, patients are followed up at 1-2 weeks and 1 month, then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed breast carcinoma or breast carcinoma in situ desiring unilateral or bilateral deep inferior epigastric perforator (DIEP) flap breast reconstruction
* Patients must be candidates for elective surgery, without clinically significant cardiac or pulmonary disease (New York Heart Association [NYHA] class III/IV), without infection requiring antibiotics, and without serious illness requiring the use of steroids
* Patients must have normal kidney function and no allergy to intravenous (IV) dye

Exclusion Criteria:

* Patients with previous abdominal donor site flaps will be excluded along with patients with previous extensive surgery to the anterior abdomen
* Patients with a weight of over 300 pounds or a body size not supported by the CT scanner will be excluded
* Patients who are expected to undergo postoperative radiation therapy will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The number of perforators that are found intraoperatively but not seen preoperatively on CT angiogram images | Up to 2 years
Whether the preoperative CT angiography allowed the surgeon to accurately predict the perforator vessels that were actually used in the final flap design and transfer | Up to 2 years

SECONDARY OUTCOMES:
Position of the vessels on the imaging correlate to actual location on the abdominal wall for those perforator vessels that are identified both on preoperative review of the images and located during flap dissection | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Kocak, MD, Principal Investigator — Ohio State University

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu